CLINICAL TRIAL: NCT04901052
Title: Effect of a Diet Supplemented with Omega-3 on Biochemical Variables, Cytokine Concentration and Fatty Acid Profile in Subjects with Obesity
Brief Title: Effects of N-3 Intake on Lipid Profile, Biochemical and Inflammatory Markers in Subjects with Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Centro Universitario de Ciencias de la Salud, Mexico (Other); Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-01219
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2021-05

CONDITIONS: Obesity
Keywords: Dietary Supplementations; Anti-Inflammatory Agent
MeSH Terms: conditions — Obesity | interventions — Sunflower Oil

STUDY DESIGN:
Intervention Model Description: Randomized Parallel with placebo
Who Masked: Participant, Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- n-3 supplementation group (Experimental): The nutritional strategy consisted a hypocaloric diet high in n-3. A 20% reduction by the total estimated energy through the Mifflin-St.Jeor formula was calculated, following a 50% to carbohydrates, 20% to proteins and 30% to lipids distribution. All participants received a balanced nutritional plan of omega-6/omega-3 close to 5:1 ratio, according to estimated energy. Additionally, a high omega-3 foods list was proportioned to emphasize their consumption during the study plus Omega 3 supplementation, the dosage was 2 capsules per day, containing 1.5 g of omega 3, of which 1000 mg were EPA and 500mg DHA. The omega 3 capsules were obtained from the same batch.
  Interventions: Dietary Supplement: n-3 supplementation group
- Placebo group (Placebo Comparator): The nutritional strategy consisted a hypocaloric diet high in n-3. A 20% reduction by the total estimated energy through the Mifflin-St.Jeor formula was calculated, following a 50% to carbohydrates, 20% to proteins and 30% to lipids distribution. All participants received a balanced nutritional plan of omega-6/omega-3 close to 5:1 ratio, according to estimated energy. Additionally, a high omega-3 foods list was proportioned to emphasize their consumption during the study plus placebo capsules (2 capsules per day made from sunflower oil)
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: n-3 supplementation group — n-3 supplementation group (1.5g of omega 3)
  Arms: n-3 supplementation group
Dietary Supplement: Placebo group — Placebo group (sunflower oil)
  Other Names: Placebo group (sunflower oil)
  Arms: Placebo group

SUMMARY:
Obesity is a chronic disease characterized by the excessive accumulation of adipose tissue that is harmful to health. Dietary habits modification through a caloric restriction, macronutrient distribution including linoleic and linolenic (n-6:n-3) polyunsaturated fatty acids (PUFAs) ratio, has been suggested for obesity management. It has been proposed that the optimal n-6: n-3 ratio should be between 1:1 and 5:1 to maintain a healthy balance. Purpose: Compare the effect of a diet n6:n3 ratio of polyunsaturated fatty acids with a group supplemented with n-3 PUFA on lipid profile in erythrocyte membrane, biochemical and inflammatory markers in subjects with obesity.

Methods: 58 subjects were randomly divided into two groups: fish oil group and the placebo group. Anthropometric and biochemical data were evaluated, cytokine levels was performed using the Bio-PlexPro™ HumanTh17Cytokine Assays (MagPix) panel. The fatty acid profile quantification in the erythrocyte membrane was carried out by gas chromatography. Statistical analysis was performed with Statistical Package for the Social Sciences (SPSS) v.22 software.

DETAILED DESCRIPTION:
A randomized clinical trial was conducted at the Institute of Translational Nutrigenetics and Nutrigenomics of the University of Guadalajara. All participants were recruited through flyers and social media invitations. Sample size was determined according to the mean difference formula for clinical trials. To achieve a statistical power of 80% and an alpha of 5%, a sample size of 19 participants in each study group was required. However, 58 obese individuals who met the selection criteria were randomized in n-3 group or placebo group.

Blood sample, height and weight were measured after 8-12 hour fast and wearing light clothes.

The nutritional intervention consisted in 20% reduction by the total estimated energy through the Mifflin-St.Jeor formula was calculated, following a 50% to carbohydrates, 20% to proteins and 30% to lipids distribution. All participants received a balanced nutritional plan of omega-6/omega-3 close to 5:1 ratio, according to estimated energy. Additionally, a high omega-3 foods list was proportioned to emphasize their consumption during the study. Fish oil group besides the diet was supplemented with omega 3, the dosage was 2 capsules per day, containing 1.5 g of total omega 3, of which 1000 mg were EPA and 500mg DHA. The omega 3 capsules were obtained from the same batch, and a toxicity analysis was performed to verify the safety or the placebo group (2 capsules per day made from sunflower oil).

This study was approved by the Ethics and Biosafety Committee of the Health Sciences Center, University of Guadalajara (Registration number CI-01219) and was carried out according to the Declaration of Helsinki (2013) and all the participants signed a written consent-informed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes
* Mestizo from West Mexico
* Age between 30 to 50 years of age
* Sign the Informed Consent
* Diagnostic of Obesity type I and II according to BMI (30 - 40kg / m2)
* Waist circumference (WC) women ≥80cm, men ≥90cm
* Sedentary lifestyle ˂ 150 minutes per week

Exclusion Criteria:

* Pregnant or breastfeeding women
* Diabetes disease
* Cardiovascular disease
* Any type of cancer disease Tobacco and alcohol (consumption ≥ 40 g of alcohol per day for men and ≥ 20 g for women)
* Participants that consume n-3 supplements, anti-inflammatory medications, or some type of lipid-lowering drugs in the past year

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
The fatty acid profile quantification | Mean change from baseline (0 Month) to end of treatment at 4th Month
  All the samples was performed in a Gas Chromatograph (GC) Agilent Technologies, 6850 network system coupled to an injector (Agilent Technologies, 7083 Series) with a column for fatty acids (Durabond, DB-23). flame ionization detector with helium as gas carrier (0.7 cm3 min-1) and a temperature ramp (110 °C - 220 °C).
Pro-inflammatory and Anti-inflammatory Cytokines profile in serum | Mean change from baseline (0 Month) to end of treatment at 4th Month
  The pro-inflammatory and anti-inflammatory cytokines quantification were using Bio-Plex Pro™ Human cytokine Standard 17-Plex, Group I kit following the supplier's instructions, and the read was immediately by MAGPIX™ analyzer.
  The 17 cytokine include: IL1β, IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL17A, G-CSF, GM-CSF, INF-γ, MCP-1, MIP1α, TNFα. Units of measure in pg/ml.

SECONDARY OUTCOMES:
Changes in Weight | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  The weight was measured in kilograms on InBody 370
Changes in Body Mass Index (BMI) | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  Weight and height were be combined to report BMI in kg/m^2
Changes in Waist Circumference | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month.
  Waist circumference was measured at the narrowest point between the edge of the inner rib and the iliac crest, with the participant in an abducted and relaxed position, after expiration using a Lufkin Executive® tape.
Changes in Fat Mass | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  The Fat Mass was measured in kilograms by electrical bioimpedance on InBody 370.
Changes in Serum Glucose | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Serum Insulin | At the baseline (0 Month) and the 4th month
  Were determined through Insulin Model ELISA kit following the supplier's instructions.
Changes in homeostatic model assessment - insulin resistance (HOMA-IR) | At the baseline (0 Month) and the 4th month
  Serum glucose and Insulin levels were be combined to report HOMA-IR calculated as described by Matthews.
Changes in Total Cholesterol | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in High-density lipoprotein (c-HDL) | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  It was measured in mg/dL using a dry chemistry system in Vitros 350 equipment.
Changes in Low-density lipoprotein (c-LDL) | At the baseline (0 Month) and 1st month, 2nd month, 3th month and the 4th month
  It was calculated using Friedewald formula

CONTACTS AND LOCATIONS:
Overall Officials: Erika Martinez-Lopez, PhD, Study Director — University of Guadalajara
Locations (2):
- Mexico (2):
  - University of Guadalajara, Guadalajara, Jaliscco
  - Erika Martínez-López, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared to protect and safeguard the confidentiality data of the participants.

REFERENCES:
- [Background] Albracht-Schulte K, Kalupahana NS, Ramalingam L, Wang S, Rahman SM, Robert-McComb J, Moustaid-Moussa N. Omega-3 fatty acids in obesity and metabolic syndrome: a mechanistic update. J Nutr Biochem. 2018 Aug;58:1-16. doi: 10.1016/j.jnutbio.2018.02.012. Epub 2018 Feb 27. PMID 29621669
- [Background] Torres-Castillo N, Silva-Gomez JA, Campos-Perez W, Barron-Cabrera E, Hernandez-Canaveral I, Garcia-Cazarin M, Marquez-Sandoval Y, Gonzalez-Becerra K, Barron-Gallardo C, Martinez-Lopez E. High Dietary omega-6:omega-3 PUFA Ratio Is Positively Associated with Excessive Adiposity and Waist Circumference. Obes Facts. 2018;11(4):344-353. doi: 10.1159/000492116. Epub 2018 Aug 10. PMID 30092569
- [Background] Vannice G, Rasmussen H. Position of the academy of nutrition and dietetics: dietary fatty acids for healthy adults. J Acad Nutr Diet. 2014 Jan;114(1):136-53. doi: 10.1016/j.jand.2013.11.001. PMID 24342605
- [Background] Bruun JM, Lihn AS, Madan AK, Pedersen SB, Schiott KM, Fain JN, Richelsen B. Higher production of IL-8 in visceral vs. subcutaneous adipose tissue. Implication of nonadipose cells in adipose tissue. Am J Physiol Endocrinol Metab. 2004 Jan;286(1):E8-13. doi: 10.1152/ajpendo.00269.2003. Epub 2003 Sep 16. PMID 13129857
- [Background] Oh DY, Talukdar S, Bae EJ, Imamura T, Morinaga H, Fan W, Li P, Lu WJ, Watkins SM, Olefsky JM. GPR120 is an omega-3 fatty acid receptor mediating potent anti-inflammatory and insulin-sensitizing effects. Cell. 2010 Sep 3;142(5):687-98. doi: 10.1016/j.cell.2010.07.041. PMID 20813258
- [Background] Gurzell EA, Wiesinger JA, Morkam C, Hemmrich S, Harris WS, Fenton JI. Is the omega-3 index a valid marker of intestinal membrane phospholipid EPA+DHA content? Prostaglandins Leukot Essent Fatty Acids. 2014 Sep;91(3):87-96. doi: 10.1016/j.plefa.2014.04.001. Epub 2014 Apr 24. PMID 24913088
- See also: World Health Organization — https://www.who.int/es/news-room/fact-sheets/detail/obesity-and-overweight